CLINICAL TRIAL: NCT00582972
Title: Does Omeprazole Decrease Intestinal Calcium Absorption?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: H-2007-0179; 07-1235-03
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Osteoporosis; Achlorhydria; GERD; Hip Fracture
Keywords: Calcium Absorption; Fractional Calcium Absorption; Omeprazole; Stable Calcium Isotopes; Proton Pump Inhibitor; Intestinal Absorption of Calcium
MeSH Terms: conditions — Osteoporosis; Achlorhydria; Gastroesophageal Reflux; Hip Fractures | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Subjects will receive omeprazole 40 mg daily for 30 days
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — 40 mg po qAM one-half hour before breakfast for 30 days
  Other Names: Losec; Prilosec

SUMMARY:
The purpose of this study is to measure the effect of omeprazole on intestinal calcium absorption in postmenopausal women.

DETAILED DESCRIPTION:
Existing literature makes it unclear whether proton pump inhibitor therapy truly decreases intestinal calcium absorption. Up to 25 postmenopausal women will participate in this study. The primary study outcome is the change in intestinal calcium absorption following omeprazole therapy 40 mg daily for 30 days. The secondary outcomes include the change in urine n-telopeptide.

We will interview women and review their medical records to determine eligibility. Eligible subjects will undergo three calcium absorption studies. The first 2 studies will determine the monthly variation in calcium absorption, while the 3rd study will occur after taking 40 mg of omeprazole daily for 30 days. Women will present to the research unit in the early morning and receive an oral and intravenous calcium tracer with breakfast. Over the next 24 hours, we will collect all urine for measurement of its calcium content. During the first stay, we will measure each subject's gastric pH by collecting gastric fluid from a temporary nasogastric tube. In consenting subjects we will collect one tube of blood, isolate its DNA.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 5 years past menopause, defined as the last date of menses

Exclusion Criteria:

* Allergy/Intolerance to orange juice
* Allergy/Intolerance to omeprazole or other PPI therapy
* Use of drugs that interact with omeprazole including oral anti-fungal agents, coumadin, diazepam, phenytoin & tacrolimus
* Use of antacids, PPI or H2-blocker therapy within the past two months
* Intestinal conditions associated with malabsorption or low gastric acid levels including Crohn's Disease, ulcerative colitis, pernicious anemia, bacterial overgrowth, celiac sprue, chronic diarrhea or use of antibiotics within the past month
* Known Stage 4 or 5 Chronic Kidney Disease, defined as an estimated GFR <30 cc/minute
* Use of medications known to interfere with calcium metabolism, including oral steroids or anticonvulsants

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Hansen, MD, Principal Investigator — Univeristy of Wisconsin School of Medicine and Public Health
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Hansen KE, Jones AN, Lindstrom MJ, Davis LA, Ziegler TE, Penniston KL, Alvig AL, Shafer MM. Do proton pump inhibitors decrease calcium absorption? J Bone Miner Res. 2010 Dec;25(12):2786-95. doi: 10.1002/jbmr.166. Epub 2010 Jun 24. PMID 20578215
- [Result] Jones AN, Shafer MM, Keuler NS, Crone EM, Hansen KE. Fasting and postprandial spot urine calcium-to-creatinine ratios do not detect hypercalciuria. Osteoporos Int. 2012 Feb;23(2):553-62. doi: 10.1007/s00198-011-1580-7. Epub 2011 Feb 24. PMID 21347742

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At least 5 years past onset of menopause; not taking proton pump inhibitors
Pre-assignment Details: subjects completed a food diary
Period: Overall Study
Arm/Group | Experimental
Started | 23
Completed | 21
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Intestinal Calcium Absorption From Baseline to One Month
Description: percent calcium absorption
Time Frame: change in calcium absorption from baseline to 1 month
Population: Subjects completing the measures of calcium absorption were included in the analysis of the primary outcome.
Measure: Mean (Standard Deviation); unit: percent calcium absorption
Groups:
- Experimental: omeprazole 40 mg daily for 30 days
Arm/Group | Experimental
Number analyzed (Participants) | 21
percent calcium absorption | 5 (10)

2. Secondary Outcome: Change in Bone Resorption From Baseline to 1 Month
Description: urine n-telopeptide (normalized to creatinine levels)
Time Frame: change in bone resorption from baseline to 1 month
Population: 23 enrolled but two dropped from the study, leading to 21 subjects who completed all study visits
Measure: Mean (Standard Deviation); unit: mcg/mmol creatinine
Groups:
- Experimental: Subjects received omeprazole 40 mg daily for 30 days
Arm/Group | Experimental
Number analyzed (Participants) | 21
mcg/mmol creatinine | 1.9 (0.9)

ADVERSE EVENTS:
Arm/Group | Experimental
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No